CLINICAL TRIAL: NCT04567888
Title: Testing a Digital Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happify Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HLS-20
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Rumination; Stress, Psychological
MeSH Terms: conditions — Rumination Syndrome; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Users are randomly assigned between arms after completing baseline assessment and stay in that arm for the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Happify Teens (Active Comparator): Happify Teens is a digital well-being intervention that can be accessed via mobile application or web browser
  Interventions: Behavioral: Happify Teens
- Waitlist Control (No Intervention): Waitlist Control Condition

INTERVENTIONS:
Behavioral: Happify Teens — An online platform for conveying techniques from positive psychology, cognitive-behavioral therapy, and mindfulness-based stress reduction.
  Arms: Happify Teens

SUMMARY:
Teen participants (ages 13-17) will be randomly assigned to either an experimental (the Happify Teens digital platform), or a waitlist control group. The study includes an 8-week intervention period and a 1-month follow up period.

DETAILED DESCRIPTION:
Teen participants (ages 13-17) will be randomly assigned to either the experimental group in which participants receive access to Happify Teens, a digital platform rooted in several therapeutic traditions that aims to improve wellbeing, or a waitlist control group. Both group conditions last 8 weeks. Participants assigned to the Happify Teens platform will have full access to the intervention, with featured tracks that focus on dealing with stress, worries and building skills for greater happiness. Participants assigned to the waitlist (control) condition will not have access to the Happify Teens platform for the full study period (12 weeks total). Participants in the waitlist control will receive access to Happify Teens after the full study period is complete (12 weeks). Perceived stress, rumination, and optimism will be assessed via self-report at baseline, end of the 8-week intervention, and at 1 month post intervention.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years of age
* US resident
* Perceived Stress Scale Score ≥ 10
* Ruminative Responses Scale Score ≥ 14
* Ability and willingness to complete study activities
* Willingness and access to using a digital intervention via mobile application or web browser

Exclusion Criteria:

* Current or past user of any Happify platform
* Non-US Resident
* Perceived Stress Scale Score < 10
* Ruminative Responses Scale Score < 14

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 353 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Boucher, PhD, Principal Investigator — Happify Inc.
Locations (1):
- Happify (an online platform -- study is entirely online), New York, New York, United States

REFERENCES:
- [Derived] Boucher EM, Ward H, Miles CJ, Henry RD, Stoeckl SE. Effects of a Digital Mental Health Intervention on Perceived Stress and Rumination in Adolescents Aged 13 to 17 Years: Randomized Controlled Trial. J Med Internet Res. 2024 Mar 29;26:e54282. doi: 10.2196/54282. PMID 38551617
- [Derived] Boucher EM, Ward HE, Stafford JL, Parks AC. Effects of a Digital Mental Health Program on Perceived Stress in Adolescents Aged 13-17 Years: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Apr 19;10(4):e25545. doi: 10.2196/25545. PMID 33871377

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Happify Teens | Waitlist Control
Started | 178 | 175
Completed | 132 | 171
Not Completed | 46 | 4
Not completed — Did Not Create Happify for Teens Account | 22 | 0
Not completed — Did Not Complete Any Happify for Teens Activities | 22 | 0
Not completed — Reported Unusual Birth Year | 2 | 3
Not completed — Duplicate Responses | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Happify Teens | Waitlist Control | Total
Number analyzed (Participants) | 178 | 175 | 353
Age, Customized [Count of Participants; unit: Participants]
  13 years | 19 | 24 | 43
  14 years | 44 | 42 | 86
  15 years | 30 | 31 | 61
  16 years | 36 | 43 | 79
  17 years | 47 | 32 | 79
  Missing or Unusual Birth Year | 2 | 3 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 122 | 110 | 232
  Male | 42 | 50 | 92
  Non-Binary/Other | 14 | 14 | 28
  Missing | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 22 | 41
  Not Hispanic or Latino | 159 | 153 | 312
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 140 | 138 | 278
  More than one race | 17 | 15 | 32
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 178 | 175 | 353
Perceived Stress Scale [Mean (Standard Deviation); unit: score on a scale] — 10-item measure of perceived stress scoring how often the participant felt stressed by each statement in the following month from never (0) to very often (4). Scores can range from 0 to 40, with higher scores indicating higher levels of perceived stress.
  score on a scale | 26.06 (4.41) | 25.29 (5.04) | 25.68 (4.74)
Ruminative Responses Scale - Brooding Subscale [Mean (Standard Deviation); unit: score on a scale] — A 5-item measure of rumination (brooding) scoring how often participants engage with each of the 5 behaviors on a scale from almost never (1) to almost always (4). Ratings are summed, so that total scores can range from 5 to 20, with higher scores indicating more brooding in the past month.
  score on a scale | 14.18 (2.32) | 14.29 (2.55) | 14.23 (2.44)

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress [Perceived Stress Scale (PSS)]
Description: 10-item measure of perceived stress scoring how often the participant felt stressed by each statement in the following month from never (0) to very often (4). Scores can range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Happify Teens | Waitlist Control
Number analyzed (Participants) | 132 | 171
score on a scale
  Baseline | 26.33 (4.43) | 25.26 (4.97)
  4 weeks | 22.01 (6.10) | 24.67 (5.36)
  8 weeks | 21.95 (6.20) | 24.61 (6.10)
  12 weeks | 20.96 (6.57) | 24.44 (6.27)
Statistical Analysis 1: Comparison: Happify Teens vs Waitlist Control; Test type: Superiority; p < .001, Repeated-measures Multilevel Models — Threshold for statistical significance set to .050; Slope = -1.41, 95% CI 2-sided [-1.88 to -0.95]

2. Secondary Outcome: Change in Rumination [Ruminative Responses Scale (RRS)-Short Form-Brooding Subscale]
Description: A 5-item measure of rumination (brooding) assessing how often participants engage with each of the 5 behaviors on a scale from almost never (1) to almost always (4). Ratings are summed so that total scores can range from 5 to 20, with higher scores indicating more brooding in the past month.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Happify Teens | Waitlist Control
Number analyzed (Participants) | 132 | 171
score on a scale
  Baseline | 14.29 (2.36) | 14.29 (2.56)
  4 weeks | 12.53 (3.24) | 13.89 (3.01)
  8 weeks | 11.94 (2.89) | 13.20 (2.85)
  12 weeks | 11.68 (3.18) | 13.46 (3.03)
Statistical Analysis 1: Comparison: Happify Teens vs Waitlist Control; Test type: Superiority; p < .001, Repeated-measures Multilevel Models — Threshold for statistical significance was set to .050; Slope = -0.54, 95% CI 2-sided [-0.78 to -0.30]

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Happify Teens | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04567888/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04567888/SAP_001.pdf